CLINICAL TRIAL: NCT05235828
Title: Sudarshan Kriya Yoga for Canadian Veterans With Post-Traumatic Stress Disorder: A Nation-wide Effectiveness and Implementation Evaluation
Brief Title: Studying the Effectiveness and Implementation of Sudarshan Kriya Yoga for Canadian Veterans With PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Atlas Institute for Veterans and Families (Unknown); St. Joseph's Health Care London (Other); Quebec City Operational Stress Injury Clinic (Unknown); Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ross Upshur, Physician researcher, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 21-0275-A
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: PTSD; Depressive Symptoms; Anxiety; Pain; Quality of Life; Post Traumatic Stress Disorder
Keywords: Veteran; Armed forces; Royal Canadian Mounted Police; RCMP; Meditation; Sudarshan Kriya Yoga; Breathing-based meditation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Waitlist control design with an active intervention (ACT) and waitlist control (WLC) group. The ACT group will receive the v-SKY intervention after the baseline assessment while the WLC group will have a 6-week waitlist period. Afterwards, the WLC group will receive the v-SKY intervention while the other group will receive no intervention for 6 weeks.
Who Masked: Outcomes Assessor
Masking Description: The member of the research team who is assessing outcome measures will be blinded to the randomization outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (ACT) group (Experimental): 8-12 participants will meet for 3-hour sessions for the first 5 days of the intervention. This is followed by five weeks of 1-hour sessions twice per week. In total, the intervention will be 15 sessions that run for a total of 25 hours over 6-weeks. Experienced and licensed SKY instructors from the International Association for Human Values (IAHV) and Art of Living Foundation (AOLF) will provide the intervention through video calls. Instructors will guide participants through the v-SKY intervention through visual demonstrations and verbal guidance. All sessions will be delivered virtually using Zoom. Sessions will not be recorded.
  Interventions: Behavioral: Sudarshan Kriya Yoga (SKY)
- Waitlist control (WLC) group (No Intervention): 8-12 participants will not receive the intervention for 6-weeks. The 6-weeks will line up with the v-SKY intervention that the ACT group receives. After the waitlist period, the WLC group will receive the same v-SKY intervention as the ACT group. According to our earlier estimates, a high number of veterans with PTSD may not be actively receiving treatment for their illness. For these reasons, a waitlist control design may better reflect the current treatment environment for veterans with PTSD.

INTERVENTIONS:
Behavioral: Sudarshan Kriya Yoga (SKY) — This is the experimental arm of the study, where participants will be trained in a form of breathing based meditation that incorporates different breathing techniques centred around controlling arousal and attention. Participants will be encouraged to learn all of the techniques that are covered during these sessions and also utilize the techniques that are most appropriate for their personal needs. After some initial training sessions, participants will be encouraged to practice their new SKY techniques in environments and situations that they have been avoiding. They would begin with situations that are less triggering, and progress to more difficult situations. At each group session, participants will describe their experiences and discuss ways to continue to incorporate the SKY techniques into their daily lives, until it reaches a point of being natural to use these skills throughout the day, both in practice, and in application.
  Arms: Active intervention (ACT) group

SUMMARY:
We plan to study the reach, effectiveness, adoption, implementation, and maintenance of the virtually-delivered Sudarshan Kriya Yoga (v-SKY) intervention. We will study effectiveness by comparing the effects of v-SKY to a waitlist control in a randomized controlled trial (RCT) with Canadian military and RCMP veterans with PTSD. Effects of the intervention on PTSD symptom severity, depression, pain, anxiety, and quality of life will be evaluated. We will evaluate the reach, adoption, implementation, and maintenance of the v-SKY intervention amongst veterans, SKY instructors, health professionals, and administrators by interviewing RCT participants, instructors, health professionals, and administrators that work with veterans. Evaluating implementation of a virtual intervention is relevant in both pandemic and post-pandemic contexts where virtual interventions may continue to be more available and possibly preferred by patients and clients.

DETAILED DESCRIPTION:
Using a mixed-methods approach guided by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, we will conduct a hybrid type II effectiveness/implementation study1 consisting of a randomized controlled trial (RCT) and a parallel implementation evaluation of Sudarshan Kriya Yoga for Canadian veterans.

OBJECTIVES:

To determine the effect of v-SKY on decreasing PTSD symptom severity, quality of life, and depressive, anxiety, and pain symptoms in Canadian veterans affected by PTSD.

To evaluate the implementation of the v-SKY intervention amongst Canadian veterans with PTSD and the health professionals, and administrators that work with veterans, by evaluating the reach, adoption, implementation, and maintenance of the intervention.

RCT RECRUITMENT AND CONSENT: Participants who are veterans of the Canadian Armed Forces (CAF) or Royal Canadian Mounted Police (RCMP) with PTSD will be recruited through various organizations and clinics across Canada. All potential participants will be provided with a consent form and given as much time as needed to consider participation. After this time, informed consent will be obtained from those interested in participating and they will be screened for eligibility by study staff.

STUDY INTERVENTION: SKY meditation is a standardized intervention that includes relaxation techniques as well as periods of group discussion. It will be taught over Zoom by trained and certified teachers from the International Association of Human Values (IAHV) and Art of Living Foundation (AOLF). Groups of 8-12 Canadian veterans will be taught the SKY intervention over a 6-week period. Raters and instructors will be blind to participant's randomization outcome. Half of the participants will receive the v-SKY intervention within 2-weeks of the baseline assessment while the other half will receive the v-SKY intervention after a 6-week waitlist period.

DATA COLLECTION: Participants will be screened for eligibility using the PTSD Checklist for DSM-5 (PCL-5) and Mini International Neuropsychiatric Interview Screen and Standard 7.0.2 (MINI). The primary outcome (PTSD symptom severity) will be evaluated using the PCL-5. Exploratory outcomes (quality of life and symptoms of depression, anxiety, and pain) will be evaluated using the Short-form 36 (SF-36), Patient Health Questionnaire-9 (PHQ-9), Generalized Anxiety Disorder scale (GAD-7), and Brief Pain Inventory (BPI), respectively. Measures of primary and exploratory outcomes will be administered at all 4 assessment sessions and are described below:

At the baseline assessment the following information will be collected:

Intake survey that will collect demographic information on age, partial date of birth (DOB), gender, ethnicity, employment status, military and/or RCMP service status, housing type, household finances, highest level of education achieved, smoking, caffeine intake, drug and alcohol use, duration of PTSD diagnosis, and past treatment history for their PTSD. Participants will also be asked about their psychiatric history including age of first contact with services for mental illness (and which illness), history of hospital admissions and health service use.

PCL-5 [past-week version] CAPS-5 [past-month version] PHQ-9 BPI GAD-7 SF-36 Medication log collecting medication names, dosages, dosages per day, total daily dosage, and reason for use will be recorded, including vitamins and over-the-counter (OTC) medications.

During the 6-week, 12-week, and 30-week follow-up assessments the following questionnaires and measurements will be completed:

i. PCL-5, ii. PHQ-9; iii. BPI; iv. GAD-7; v. SF-36; vi. Medication log.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* CAF or RCMP veteran.
* Meet criteria for current PTSD as determined by a score of >38 on the PTSD Checklist-5 (PCL-5).

Exclusion Criteria:

* Participation in another concurrent clinical trial.
* Intention to begin a new course of Behavioural Therapy (e.g., Cognitive Behavioural Therapy including Prolonged Exposure or Cognitive Processing Therapy) during the intervention period.
* Past participation in virtual or in-person SKY.
* Initiated psychotropic medication within 8 weeks prior to the initial screening. Excluded participants could be re-considered for eligibility after stability on medication was achieved.
* Risk of imminent suicidal intent at screening as per MINI screening and standard tool. Such patients will be advised to visit their local emergency department.
* Mental disorders including schizophrenia, bipolar I, psychosis of any type.
* Seizure disorder not well controlled.
* Moderate or severe substance use disorder as per the MINI.
* Neurocognitive impairment as determined by a score of 23 or less on the Montreal Cognitive Assessment (MOCA) mini version.
* Unable to connect to the internet and use Zoom for study assessments and interventions.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms | Baseline (Week 0), Follow-up 1 (Week 6), Follow-up 2 (Week 12), Follow-up 3 (Week 30)
  The PCL-5 is a well-validated, widely used, and easy to administer 20-item self-report scale that is used in PTSD research and clinical practice. Change in PCL-5 scores from baseline to post-treatment will be measured. Prolonged effects of the interventions on PTSD symptoms will be captured with the PCL-5 at the follow-up assessments. Responses to each item relate to the four symptom clusters for PTSD, for which separate scores can be measured. These scores will be used for additional analyses.

OTHER OUTCOMES:
Change in depressive symptoms | Baseline (Week 0), Follow-up 1 (Week 6), Follow-up 2 (Week 12), Follow-up 3 (Week 30)
  PHQ-9 is a well-validated and widely used self-report scale used in depression research. Each item is rated on a 4 point scale for how much it bothered the participant in the past 2 weeks. Change in PHQ-9 scores from baseline to post-treatment will be measured. A self-report scale is more feasible than an assessor-rated scale (e.g. HAM-D17) given the virtual nature of this study. Prolonged effects of the intervention on depression symptoms will be captured with the PHQ-9 at the follow-up assessments.
Change in pain symptoms | Baseline (Week 0), Follow-up 1 (Week 6), Follow-up 2 (Week 12), Follow-up 3 (Week 30)
  The Brief pain inventory (BPI) is a validated self-report scale used in pain trials and clinical pain practice and is a core outcome measure per the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials recommendations. Two independent and clinically relevant measures are included: pain severity and pain interference with function. Change in BPI scores from baseline to post-treatment will be measured. Prolonged effects of the intervention on pain symptoms will be captured with the BPI at the follow-up assessments.
Change in anxiety symptoms | Baseline (Week 0), Follow-up 1 (Week 6), Follow-up 2 (Week 12), Follow-up 3 (Week 30)
  GAD-7 is a validated and efficient tool that is used to screen and assess the severity of GAD clinically and in research. Each of the 7-items are rated on a 4-point scale for how often it bothered the participant in the past two weeks. Change in GAD-7 scores from baseline to post-treatment will be measured. Prolonged effects of the intervention on anxiety symptoms will be captured with the GAD-7 at the follow-up assessments.
Change in quality of life | Baseline (Week 0), Follow-up 1 (Week 6), Follow-up 2 (Week 12), Follow-up 3 (Week 30)
  Change in health related quality of life (SF-36) has been validated as quality of life measurement and is recommended by IMMPACT. This measure is well-aligned to the intervention which may also improve overall quality of life in addition to specific PTSD symptom improvement. Change in SF-36 scores from baseline to post-treatment will be measured. Prolonged effects of the intervention on quality of life will be captured with the SF-36 at the follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Upshur, MD, Principal Investigator — Sinai Health System; Abhimanyu Sud, MD, Principal Investigator — Sinai Health System
Locations (1):
- Sinai Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Hoge CW, Grossman SH, Auchterlonie JL, Riviere LA, Milliken CS, Wilk JE. PTSD treatment for soldiers after combat deployment: low utilization of mental health care and reasons for dropout. Psychiatr Serv. 2014 Aug 1;65(8):997-1004. doi: 10.1176/appi.ps.201300307. PMID 24788253
- [Background] Taylor SL, Hoggatt KJ, Kligler B. Complementary and Integrated Health Approaches: What Do Veterans Use and Want. J Gen Intern Med. 2019 Jul;34(7):1192-1199. doi: 10.1007/s11606-019-04862-6. Epub 2019 Apr 22. PMID 31011973
- [Background] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Background] Carter, J. et al. Multi-component yoga breath program for Vietnam veteran post traumatic stress disorder: randomized controlled trial. J Trauma Stress Disor Treat 2 3, (2013).
- [Background] Mathersul DC, Tang JS, Schulz-Heik RJ, Avery TJ, Seppala EM, Bayley PJ. Study protocol for a non-inferiority randomised controlled trial of SKY breathing meditation versus cognitive processing therapy for PTSD among veterans. BMJ Open. 2019 Apr 3;9(4):e027150. doi: 10.1136/bmjopen-2018-027150. PMID 30948610
- [Background] Katzman MA, Vermani M, Gerbarg PL, Brown RP, Iorio C, Davis M, Cameron C, Tsirgielis D. A multicomponent yoga-based, breath intervention program as an adjunctive treatment in patients suffering from generalized anxiety disorder with or without comorbidities. Int J Yoga. 2012 Jan;5(1):57-65. doi: 10.4103/0973-6131.91716. PMID 22346068
- [Background] Hamilton-West K, Pellatt-Higgins T, Sharief F. Evaluation of a Sudarshan Kriya Yoga (SKY) based breath intervention for patients with mild-to-moderate depression and anxiety disorders. Prim Health Care Res Dev. 2019 Jun 20;20:e73. doi: 10.1017/S1463423619000045. PMID 32799993
- [Background] Vasudev K, Ionson E, Inam S, Speechley M, Chaudhari S, Ghodasara S, Newman RI, Vasudev A. Sudarshan Kriya Yoga Program in Posttraumatic Stress Disorder: A Feasibility Study. Int J Yoga. 2020 Sep-Dec;13(3):239-246. doi: 10.4103/ijoy.IJOY_16_20. Epub 2020 Sep 13. PMID 33343155